CLINICAL TRIAL: NCT00735514
Title: Adherence to Vaginal Dilation Following Pelvic Radiotherapy for Gynecological Cancers
Brief Title: Compliance to Vaginal Dilation Therapy in Patients Who Have Undergone Radiation Therapy For Stage IB, Stage IIA, Stage IIB, Stage IIIA, or Stage IIIB Cervical Cancer or Stage IA, Stage IB, Stage IIA, or Stage IIB Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE5808; P30CA043703 (NIH); CASE5808 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Cervical Cancer; Endometrial Cancer; Radiation Toxicity; Sexuality and Reproductive Issues
Keywords: radiation toxicity; sexuality and reproductive issues; stage I endometrial carcinoma; stage II endometrial carcinoma; stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; stage III cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Radiation Injuries; Sexuality | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: compliance monitoring — Patients from the IMPAC registry in Radiation Oncology at the University Hospitals Case Medical Center, Ireland Cancer Center complete questionnaires online or by mail. Questionnaires include the Vaginal Dilation Adherence questionnaire, the Sexual Function-Vaginal Changes Questionnaire, the Dyadic Satisfaction questionnaire, and the Physician/Nurse Recommendation of Vaginal Dilation questionnaire.
Other: questionnaire administration — Patients from the IMPAC registry in Radiation Oncology at the University Hospitals Case Medical Center, Ireland Cancer Center complete questionnaires online or by mail. Questionnaires include the Vaginal Dilation Adherence questionnaire, the Sexual Function-Vaginal Changes Questionnaire, the Dyadic Satisfaction questionnaire, and the Physician/Nurse Recommendation of Vaginal Dilation questionnaire.
Procedure: assessment of therapy complications — Patients from the IMPAC registry in Radiation Oncology at the University Hospitals Case Medical Center, Ireland Cancer Center complete questionnaires online or by mail. Questionnaires include the Vaginal Dilation Adherence questionnaire, the Sexual Function-Vaginal Changes Questionnaire, the Dyadic Satisfaction questionnaire, and the Physician/Nurse Recommendation of Vaginal Dilation questionnaire.
Procedure: management of therapy complications — Patients from the IMPAC registry in Radiation Oncology at the University Hospitals Case Medical Center, Ireland Cancer Center complete questionnaires online or by mail. Questionnaires include the Vaginal Dilation Adherence questionnaire, the Sexual Function-Vaginal Changes Questionnaire, the Dyadic Satisfaction questionnaire, and the Physician/Nurse Recommendation of Vaginal Dilation questionnaire.
Procedure: psychosocial assessment and care — Patients from the IMPAC registry in Radiation Oncology at the University Hospitals Case Medical Center, Ireland Cancer Center complete questionnaires online or by mail. Questionnaires include the Vaginal Dilation Adherence questionnaire, the Sexual Function-Vaginal Changes Questionnaire, the Dyadic Satisfaction questionnaire, and the Physician/Nurse Recommendation of Vaginal Dilation questionnaire.

SUMMARY:
RATIONALE: Understanding how well patients comply with their treatment regimen may help doctors determine best treatment and ongoing care for future patients.

PURPOSE: This phase I study is looking at compliance with vaginal dilation therapy in women who have undergone radiation therapy for stage IB, stage IIA, stage IIB, stage IIIA, or stage IIIB cervical cancer or stage IA, stage IB, stage IIA, or stage IIB endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine adherence to vaginal dilation therapy after radiotherapy in patients with early-stage IB grade 2-IIIB cervical cancer or stage IA grade 3-IIB endometrial cancer.
* To identify demographic, medical, and psychosocial factors associated with adherence to recommendations for vaginal dilation in these patients.
* To describe the sexual, marital, and non-marital dyadic functioning of these patients.

OUTLINE: Patients from the IMPAC registry in Radiation Oncology at the University Hospitals Case Medical Center, Ireland Cancer Center complete questionnaires online or by mail. Questionnaires include the Vaginal Dilation Adherence questionnaire, the Sexual Function-Vaginal Changes Questionnaire, the Dyadic Satisfaction questionnaire, and the Physician/Nurse Recommendation of Vaginal Dilation questionnaire.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* History of early-stage IB grade 2-IIIB cervical cancer or stage IA grade 3-IIB endometrial cancer
* Meets the following criteria:

  * Received radiotherapy for this disease
  * Treated within the last 3 years and followed for at least 6 months

PATIENT CHARACTERISTICS:

* Able to read and understand English
* Currently with or without a sexual partner
* No history of other cancers
* No other potentially life-threatening disease

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2008-07; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Adherence to vaginal dilation therapy after radiotherapy as measured by the Vaginal Dilation Adherence questionnaire | one time questionaire
Demographic, medical, & psychosocial factors assoc. with adherence to vaginal dilation by Vaginal Dilation Adherence questionnaire, Sexual Function-Vaginal Changes Questionnaire, & Physician/Nurse Recommendation of Vaginal Dilation questionnaire | one time questionaire
Sexual, marital, and non-marital dyadic functioning as measured by the Sexual Function-Vaginal Changes Questionnaire and the Dyadic Satisfaction questionnaire | one time questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Lois C. Friedman, PhD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (8):
- United States (8):
  - Geauga Regional Hospital, Cleveland, Ohio
  - Lake/University Ireland Cancer Center, Cleveland, Ohio
  - Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - University Suburban Health Center, Cleveland, Ohio
  - UHHS Chagrin Highlands Medical Center, Cleveland, Ohio
  - Southwest General Health Center, Cleveland, Ohio
  - UHHS Westlake Medical Center, Cleveland, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Cleveland, Ohio